CLINICAL TRIAL: NCT07002619
Title: ChOlanGiography Performed Routinely Versus Selectively During Cholecystectomy: A NAtional Registry-based Randomized Controlled Trial
Acronym: COGNAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Research department, Ersta Hospital (Unknown); Södersjukhuset (Stockholm South General Hospital) (Unknown)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COGNAC
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Cholecystolithiasis; Common Bile Duct Gall Stones
Keywords: Cholecystectomy; Intraoperative cholangiography
MeSH Terms: conditions — Cholecystolithiasis; Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine cholangiography (Active Comparator): Intraoperative cholangiography attempted, regardless of anatomy and indication
  Interventions: Procedure: Routine cholangiography
- Selective cholangiography (Active Comparator): Intraoperative cholangiography attempted only in case of uncertainty regarding anatomy
  Interventions: Procedure: Selective cholangiograpy

INTERVENTIONS:
Procedure: Routine cholangiography — Intraoperative cholangiography attempted regardless of indication and anatomy
  Arms: Routine cholangiography
Procedure: Selective cholangiograpy — Intraoperative cholangiography only attempted in case of uncertainty regarding anatomy
  Arms: Selective cholangiography

SUMMARY:
Common bile duct stones (CBDS) may be asymptomatic but can cause pancreatitis, obstructive jaundice, and/or cholangitis. In Sweden, intraoperative cholangiography (IOC) is usually performed during gallstone surgery in order to detect CBDS and proactively extract them. The intervention to extract them may, however, cause complications by itself such as pancreatitis, bleeding, or perforation. In many countries, IOC is performed selectively when CBDS are suspected preoperatively (by patient history, imaging, or blood tests), or if the anatomy is unclear. There is a knowledge gap regarding the relation between risks associated with refraining from IOC and, thus, leaving undetected CBDS in situ, or actively diagnosing and removing the stones.

To compare these risks, we propose a national multicenter randomized controlled trial. The study will be embedded in the Swedish Registry for Gallstone Surgery (GallRiks), which will include all variables for inclusion and follow-up.

Population: Patients undergoing gallstone surgery without suspicion of CBDS Intervention: IOC Control: No IOC Outcome: Readmission or reintervention (Clavien-Dindo grade ≥IIIa) related to the cholecystectomy within 12 months after the operation.

A total of 6000 patients will be recruited. The results will have the potential to provide level A evidence for routines used in gallstone surgery not only in Sweden, but also internationally.

DETAILED DESCRIPTION:
ChOlanGiography performed selectively versus routinely during cholecystectomy: a NAtional registry-based randomized Controlled trial (the COGNAC trial)

Purpose and aims Cholecystectomy for symptomatic gallstone disease is one of the most common surgical procedures worldwide. Around 13 000 cholecystectomies are performed each year in Sweden (1). In addition to causing pain and inflammation of the gallbladder, gallstones may migrate through the cystic duct into the common bile duct where they can be either asymptomatic or cause complications such as biliary obstruction, cholangitis, or pancreatitis.

To diagnose common bile duct stones (CBDS), intraoperative cholangiography (IOC) can be performed during cholecystectomy. IOC also helps to verify the anatomy of the bile ducts and may, thus, reduce the risk of intraoperative bile duct injuries (2). There are several techniques available for extraction of CBDS detected at IOC, all being associated with a risk of complications such as cholangitis, pancreatitis or bleeding. Endoscopic Retrograde Cholangiopancreatography (ERCP) is the most commonly used method with reported rates of complications in 10-15% of the procedures, ranging in severity from mild to lethal (1).

Whether IOC should be performed routinely during cholecystectomy is controversial. The aim of this study is therefore to assess whether selective or routine use of IOC is superior with regards to preventing complications/morbidity after cholecystectomy.

Survey of the field There is no consensus regarding when IOC should be performed. It is uncontroversial to recommend that patients with symptoms or laboratory findings suggestive of CBDS should undergo IOC, since these could be expected to cause complications and therefore should be extracted. In addition, IOC should be performed if the anatomy of the bile ducts is unclear during the operation in order to reduce the risk of bile duct injuries.

It is however, not clear whether IOC should be performed when there is no clinical suspicion of CBDS, since it is not known how often asymptomatic CBDS will cause complications or pass spontaneously. Routine IOC, on the one hand, may lead to overtreatment of CBDS and iatrogenic complications when removing them. On the other hand, refraining from IOC in patients without symptoms suggestive of CBDS may lead to neglect of stones that could cause serious complications in the future. A report from the Swedish Agency for Health Technology Assessment and Assessment of Social Services (SBU) in 2018 concluded that there is some evidence that IOC may reduce the risk of bile duct injuries (3), but evidence regarding management of common bile duct stones detected at IOC is still lacking.

In most other countries IOC is performed only when CBDS is suspected or if the anatomy is not satisfactory exposed intraoperatively (selective IOC). The use of selective IOC is based on the assumption that the risks associated with "unnecessary" interventions to extract CBDS outweigh those associated with undetected stones. There is, however, not sufficient scientific support to create evidence-based recommendations as to whether IOC should be performed during cholecystectomy or not in order to reduce the risk of complications in patients without signs of CBDS.

Study design The study is conducted as a multicenter registry-based randomized open controlled trial. Patients undergoing cholecystectomy for gallstone disease, or gallstone-associated complications, at centers reporting to the Swedish Registry for Gallstone Surgery and ERCPs (GallRiks) comprise the source population for this trial. Patients with obstructive jaundice, cholangitis, pancreatitis or other clinical/laboratory signs of CBDS are excluded since these conditions are usually considered indications for IOC by themselves. Randomization between selective IOC and routine IOC is done immediately before the procedure by opening of sealed envelopes with computer-generated information on group allocation after the surgeon has verified eligibility for patients who have given consent to participate. All variables required to assess the primary as well as secondary outcomes are registered routinely for study patients in GallRiks.

Patients will be followed for 1 year. For all patients undergoing cholecystectomy at centers reporting to the registry, follow-up at 1 month after surgery is performed routinely (irrespective of participation in the study or not) by the local coordinator who reviews the patient records in order to register any adverse events during this period. For patients included in the study, the same follow-up is performed at 1 year after surgery as well. If there are any concerns about the clinical interpretation of postoperative adverse events, the surgeon responsible for GallRiks at the unit is consulted. SF-36 and EQ5D are completed by the patients at baseline, and at 30 days and 1 year after surgery.

Research questions It is not known whether routine IOC reduces the risk of morbidity related to previously unknown CBDS or, on the contrary, causes overdiagnosis and overtreatment of CBDS that would have passed spontaneously if left undetected. The overwhelming question of the proposed project is therefore if use of IOC is superior in terms of reducing overall morbidity associated with cholecystectomy in patients without suspected CBDS. The main hypothesis is that IOC will cause less morbidity within one year after surgery, compared to when IOC is not performed.

Several small- or medium-sized RCTs have addressed this question, without being able to reach any firm conclusion due to lack of sufficient statistical power (5). The use of selective versus routine use of IOC in relation to risk of bile duct injuries has been evaluated by SBU without being able to establish evidence for either routine (6). Importantly, the association between IOC and risk of CBDS-related morbidity was not addressed. Taken together, this question therefore still constitutes a knowledge gap. The Swedish GallRiks Register, however, provides a unique base for addressing the current research question, with some 13 000 procedures being registered each year, near complete coverage of all variables relevant for defining eligibility criteria and outcome, and a routine follow-up of all patients that may be tracked regardless of residence.

Variables and measures Primary outcome: Readmission and/or any type of surgical, endoscopic or radiological reintervention (corresponding to Clavien-Dindo grade IIIa or higher), related to the cholecystectomy within 12 months after the cholecystectomy.

Secondary outcomes

* Procedure time
* 30-day and 1-year mortality
* Any readmission
* Any adverse event
* Cumulative hospital stay (all admissions)
* Health-related quality of life assessed by SF-36 and EQ5D
* Health care costs Material: Patient selection - population, sample Patients scheduled for laparoscopic cholecystectomy at the participating centres will be asked to participate.

Eligibility criteria

* Adult population, patient age 18 years or older undergoing laparoscopic cholecystectomy Exclusion criteria
* Procedures undertaken with the primary aim of getting access to the common bile duct.
* Clinical or laboratory findings suggestive of CBDS, including obstructive jaundice or cholangitis.
* Patients not willing/capable to give informed consent Estimated sample size and power In a study based on data from GallRiks including >38 000 patients, the prevalence of CBDS in patients undergoing cholecystectomy with no preoperative suspicion of CBDS was found to be 4.9% (4). A need for re-intervention due to complications or retained CBDS within 30 days was found in 14.9 and 25.3% in patients where intraoperative measures to extract the stones were taken or not, respectively. It could therefore be assumed that the rates of complications after 30 days would be 0.7 (4.9 x 0.149) and 1.2 (4.9 x 0.253) % in the routine and selective IOC groups, respectively.

In another, so far unpublished, series from GallRiks it was found that the need for ERCP between 30 days to 12 months after cholecystectomy was 2.9% in patients undergoing IOC compared to 4.1% in patients in which IOC was not performed (5). We therefore assume that the total risk of complications with need of reintervention during the first 12 months after cholecystectomy will be 3.6 (0.7 + 2.9) % in patients randomized to IOC and 5.3 (1.2 + 4.1) % in patients where IOC is not performed. Based on the assumption that the incidence of complications is 3.6% when IOC is performed and 5.3% when this is not done, a total of 4 602 procedures would be required to reach a chance of 80% to detect a statistically significant difference at the p<0.05 level. In order to compensate for drop-outs, we plan on including 6 000 patients.

Statistical methods The two groups will be compared statistically in accordance with "intention to treat" i.e., all randomized patients are included in the analysis. Rates of readmission/reintervention (primary endpoint) will be analysed by time-to-event models (Cox regression), whereas continuous variables will be compared by mixed models. Health economic analysis will be performed by calculation of the incremental cost-effectiveness ratio (ICER), i.e. the ratio between the difference in health care costs and the difference in quality-adjusted life-years (QALYs). The generalizability of the results will be checked by comparing included patients with patients that fulfil the inclusion criteria but were not included.

References

1. Enochsson L et al. The Swedish Registry of Gallstone Surgery and ERCP (GallRiks). A nationwide registry for quality assurance of gallstone surgery. JAMA Surg. 2013 May;148(5):471-8.
2. Törnqvist B et al. Selective intraoperative cholangiography and risk of bile duct injury during cholecystectomy. Br J Surg. 2015 Jul;102(8):952-8.
3. SBU. Intraoperativ kolangiografi vid kolecystektomi. En systematisk översikt och utvärdering av medicinska, hälsoekonomiska, sociala och etiska aspekter. Stockholm: Statens beredning för medicinsk och social utvärdering (SBU); 2018. SBU-rapport nr 292. ISBN 978-91-88437-34-1.
4. Möller M et al. Natural course vs interventions to clear common bile duct stones: data from the Swedish Registry for Gallstone Surgery and Endoscopic Retrograde Cholangiopancreatography (GallRiks). JAMA Surg. 2014 Oct;149(10):1008-13.
5. Johansson E, Österberg J, Sverdén E, Enochsson L, Sandblom G. Intervention versus surveillance in patients with common bile duct stones detected by intraoperative cholangiography: a population-based registry study. Br J Surg. 2021 Dec 1;108(12):1506-1512.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cholecystectomy

Exclusion Criteria:

* Preoperative suspicion of common bile duct stone
* Pregnancy
* Age <18 years
* Preoperative suspicion of malignancy in the gallbladder or bile ducts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Reintervention within 12 months | 12 months
  Readmission and/or any type of surgical, endoscopic or radiological reintervention (corresponding to Clavien-Dindo grade 3a or higher), related to the cholecystectomy within 12 months after the cholecystectomy

SECONDARY OUTCOMES:
Procedure time | 12 hours
  Time required to complete the cholecystectomy
Mortality | One year
  Death within one year after surgery
Hospital stay | One year
  Cumulative hospital stay, including all admissions within one year after surgery
Health-related quality of life | Six months after surgery
  Health-related quality of life assessed with SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Runfors, MD, PhD, Principal Investigator — Ersta Diakoni
Locations (1):
- Ersta Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Psuedonymized data on individual participants will be available on request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025-05-25 - 2035-05-24
Access Criteria: All information will be available by request to the principal investigator
URL: https://ki.se/media/128284/download